CLINICAL TRIAL: NCT00528775
Title: A Phase II Study of Photodynamic Therapy (PDT) Using 2-[1-hexyloxyethyl]-2 Devinyl Pyropheophorbide-a (HPPH) for Treatment of Advanced Obstructing Endobronchial Lung Cancer
Brief Title: Photodynamic Therapy Using HPPH in Treating Patients With Advanced Non-Small Cell Lung Cancer That Blocks the Air Passages
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: drug cannot be prepared commercially
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000563948; RPCI-I-98707 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPPH (Experimental): Patients will receive 4 mg/m2 HPPH (given light exposure precautions) and approximately 2 days later be treated endoscopically with 150J/cm of 665 +-5nm light.
  Interventions: Drug: HPPH; Procedure: endoscopic procedure

INTERVENTIONS:
Drug: HPPH — 4 mg/m2 IV
Procedure: endoscopic procedure — Treatment with 150 joules from laser

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug, such as HPPH, that becomes active when it is exposed to a certain kind of light. When the drug is active, tumor cells are killed. This may be an effective treatment for advanced non-small cell lung cancer that blocks the air passages.

PURPOSE: This phase II trial is studying how well photodynamic therapy using HPPH works in treating patients with advanced non-small cell lung cancer that blocks the air passages.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the efficacy of photodynamic therapy (PDT) using HPPH in patients with advanced obstructing endobronchial non-small cell lung cancer.

Secondary

* To determine palliation of symptoms in patients treated with this regimen.
* To determine the amount of HPPH taken up by the obstructing endobronchial tumors in these patients.
* To determine the extent of STAT3 cross-links, which are molecular markers of immediate PDT reaction, in the obstructing tumors of these patients before and after PDT treatment.
* To determine inflammation and apoptosis in the obstructing bronchial tumors of these patients before and after PDT treatment.

OUTLINE: Patients receive HPPH IV over 1 hour on day 1. On day 3, patients undergo photodynamic therapy (PDT) comprising laser light delivered by flexible, fiberoptic fibers passed through the biopsy channel of an endoscope. Patients undergo endoscopic debridement on day 5. If viable tumor is found outside of the initial treatment area, patients may receive another dose of laser light without additional HPPH.

Patients may undergo tumor biopsies periodically during study for optional biomarker/correlative studies. Tumor tissue samples are analyzed for STAT3 cross-links by western blotting; apoptosis and inflammation biomarkers by immunohistochemistry, TUNEL, and other immunological laboratory methods; and tumor concentrations of HPPH by fluorescence emission spectroscopy.

After completion of study treatment, patients are followed at 4-6 weeks and then periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy confirmed advanced obstructing endobronchial non-small cell lung cancer

  * May have squamous cell carcinoma, adenocarcinoma, or large cell carcinoma histology
* Ineligible for or refused surgical resection
* Local endobronchial recurrence after prior surgical resection, radiotherapy, or chemotherapy allowed
* No evidence of tumor encasement of major pulmonary vessels on CT scan of the chest

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% OR ECOG PS 0-2
* WBC ≥ 4,000/mm³
* Platelet count ≥ 100,000/mm³
* Prothrombin time < 1.5 times upper limit of normal (ULN)
* Total bilirubin ≤ 2.0 mg/dL
* Creatinine ≤ 2.0 mg/dL
* Alkaline phosphatase (hepatic) ≤ 3 times ULN
* SGOT ≤ 3 times ULN
* No contraindications for bronchoscopy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after the completion of study treatment
* Patients with underlying lung disease must be judged (by the principal investigator) able to withstand mucous/debris formation at the site of treatment
* Patients who cannot breathe due to complete upper airway obstruction and who need emergency treatment to open the airway are not eligible
* No porphyria or hypersensitivity to porphyrin or porphyrin-like compounds
* No severe chronic obstructive pulmonary disease that, in the opinion of the investigator, would preclude multiple bronchoscopies
* No partial central airway obstruction from mucous/debris formation
* No high-grade upper airway obstruction of the trachea

PRIOR CONCURRENT THERAPY:

* Any type of prior therapy (e.g., chemotherapy or radiotherapy) for lung cancer allowed
* At least 4 weeks since prior and no concurrent chemotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-08; Primary Completion 2009-11 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd L. Demmy, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPPH
Started | 6
Completed | 5
Not Completed | 1
Not completed — Other not specified | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | HPPH
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Time Frame: 6 months
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | HPPH
Number analyzed (Participants) | 0

2. Secondary Outcome: Palliation of Symptoms as Assessed by the Pulmonary Symptom Scale
Time Frame: 2 months
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | HPPH
Number analyzed (Participants) | 0

3. Secondary Outcome: Photosensitizer (HPPH) Concentration in Tumor
Time Frame: 2 months
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | HPPH
Number analyzed (Participants) | 0

4. Secondary Outcome: STAT3 Cross-links as Assessed by Western Blotting
Time Frame: 2 months
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | HPPH
Number analyzed (Participants) | 0

5. Secondary Outcome: Inflammation and Apoptosis as Assessed by Immunohistochemistry
Time Frame: 2 months
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | HPPH
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | HPPH
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPPH (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Death (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Intubation complication (Injury, poisoning and procedural complications) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HPPH (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
White blood cell disorder (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin (Investigations) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes